CLINICAL TRIAL: NCT02404090
Title: Impact of the Excess Weight Loss on Mineralization Patterns of the Knee After Bariatric Operations - a Prospective CT-osteoabsorptiometry-based Study
Brief Title: Impact of the Excess Weight Loss on Mineralization Patterns of the Knee After Bariatric Operations
Acronym: CT-OAM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Marko Kraljevic (Other)
Responsible Party: Sponsor-Investigator, Marko Kraljevic, Dr. med., Spital Limmattal Schlieren
Organization: Spital Limmattal Schlieren (Other)
Other Study IDs: SLS-001
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Obesity; Weight Loss; Knee Osteoarthritis
Keywords: Obesity; Weight Loss; Knee Osteoarthritis; Subchondral Mineralization
MeSH Terms: conditions — Obesity; Weight Loss; Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: CT-osteoarbsorptiometry — Conventional CT-scan analyzed by means of a specific tool (Analyze, Mayo Clinic).

SUMMARY:
Evaluation of the subchondral mineralization plate after excess weight loss in patientes undergoing bariatric operation by means of CT-osteoabsorptiometry.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 35
* need for bariatric operation
* knee pain (VAS > 2)

Exclusion Criteria:

* malignancy
* poor compliance
* previous bariatric operation
* pregnancy
* lack of knee pain (VAC < 2)
* previous knee operation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bariatric patients with BMI > 35 kg/m2 with knee pain (VAS > 2).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-08; Primary Completion 2020-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Mineralization changes after excess weight loss? | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Urs Zingg, MD, Principal Investigator — Spital Limmattal Schlieren